CLINICAL TRIAL: NCT05081310
Title: Cryoballoon Isolation of Superior Vena Cava in Paroxysmal Atrial Fibrillation - a Randomized Study
Brief Title: Cryoballoon Isolation of Superior Vena Cava in Paroxysmal Atrial Fibrillation
Acronym: CISPAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Vedran Velagic, MD, PhD, Assistant professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVC001
Record Dates: First submitted 2021-06-07; First posted 2021-10-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vein isolation; superior vena cava isolation; cryoballoon ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVC arm (Experimental): Patients who will receive SVC isolation by the means of cryoballoon after the PVI procedure
  Interventions: Device: superior vena cava isolation
- PVI arm (Active Comparator): Patients who will receive convectional cryoballoon PVI procedure
  Interventions: Device: pulmonary vein isolation

INTERVENTIONS:
Device: superior vena cava isolation — SVC isolation by the means of cryoballoon
  Arms: SVC arm
Device: pulmonary vein isolation — conventional pulmonary vein isolation by the means of cryoballoon
  Arms: PVI arm

SUMMARY:
There is still unresolved question whether isolation of superior vena cava (SVC) in conjunction to conventional pulmonary vein isolation (PVI) improves outcomes in the treatment of paroxysmal atrial fibrillation. The investigators are conducting a randomized study to determine if SVC isolation (in addition to pulmonary vein isolation) with the cryoballoon technology can improve freedom from atrial arrhythmias in one year follow up after the ablation.

DETAILED DESCRIPTION:
Paroxysmal atrial fibrillation can be triggered by non-pulmonary vein foci, like the superior vena cava. There are some older publications showing improved result in terms of freedom from atrial tachycardias when electrical isolation of this vessel utilizing radiofrequency energy is achieved. Recent retrospective studies showed that isolation of superior vena cava by the means of cryoballoon technology is safe and feasible procedure. Furthermore, one retrospective cohort study showed improved outcomes of SVC insolation + PVI versus PVI only strategy. To our knowledge there is still no randomized data that compared SVC isolation + PVI vs PVI only strategy when using cryoballoon technology.

The investigators want to determine if SVC isolation by the means of cryoballoon technology in conjunction with PVI can improve the patients outcomes. Also, there will be focus on the safety of the procedure, especially regarding the right sided phrenic nerve palsy. The primary objective of the study is freedom from atrial arrhythmias defined by standard postprocedural monitoring by ECG and Holter monitors. The investigators are conducting a randomized study with 1:1 randomization and planning to enroll around 100 participants with 1 year follow up. One group will receive conventional cryoballoon pulmonary vein isolation, and other group will receive SVC isolation after the PVI procedure.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation scheduled for cryoballoon the ablation of atrial fibrillation (indication not related to the study)

Exclusion Criteria:

persistent atrial fibrillation

* renal failure
* contrast allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
efficacy | one year
  number of patients free of any atrial arrhythmias during the one year of follow up (occurrence of any atrial arrhythmia longer than 30 seconds, detected by Holter EKG or 12 lead EKG will be considered as treatment failure)

SECONDARY OUTCOMES:
feasibility | during the procedure
  the success rates of SVC isolation. percentage of patients in whom successful SVC isolation was performed. SVC isolation will be verified by the circular mapping catheter, after the application of cryoballoon lesion. The absence of electrical signals in SVC after the ablation is considered as a successful isolation.
safety | one year
  adverse events during the procedure (specials consideration on phrenic nerve palsy) and after the procedure (groin hematoma, pericardial effusion, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Velagic, MD, PhD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- KBC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Overeinder I, Osorio TG, Calburean PA, Bisignani A, Bala G, Sieira J, Stroker E, Al Houssari M, Mojica J, Boveda S, Paparella G, Brugada P, de Asmundis C, Chierchia GB. Comparison between superior vena cava ablation in addition to pulmonary vein isolation and standard pulmonary vein isolation in patients with paroxysmal atrial fibrillation with the cryoballoon technique. J Interv Card Electrophysiol. 2021 Dec;62(3):579-586. doi: 10.1007/s10840-020-00932-6. Epub 2021 Jan 15. PMID 33447964
- [Background] Wei HQ, Guo XG, Sun Q, Yang JD, Xie HY, Cao ZJ, Chen YQ, Zhang S, Wu S, Ma J. Electrical isolation of the superior vena cava using second-generation cryoballoon in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2020 Jun;31(6):1307-1314. doi: 10.1111/jce.14477. Epub 2020 Apr 11. PMID 32250512
- [Background] Iacopino S, Osorio TG, Filannino P, Artale P, Sieira J, Stroker E, Bala G, Overeinder I, Hacioglu E, Calburean PA, Paparella G, Brugada P, de Asmundis C, Chierchia GB. Safety and feasibility of electrical isolation of the superior vena cava in addition to pulmonary vein ablation for paroxysmal atrial fibrillation using the cryoballoon: lessons from a prospective study. J Interv Card Electrophysiol. 2021 Mar;60(2):255-260. doi: 10.1007/s10840-020-00740-y. Epub 2020 Apr 6. PMID 32253600